CLINICAL TRIAL: NCT01609088
Title: Pilot Study of the Effects of Erythritol on Endothelial Function in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Cargill (Industry)
Responsible Party: Principal Investigator, Joseph A. Vita, Professor of Medicine, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-31447
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: endothelium; diabetes mellitus; oxidative stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erythritol-containing beverage (Experimental)
  Interventions: Dietary Supplement: Erythritol-containing beverage

INTERVENTIONS:
Dietary Supplement: Erythritol-containing beverage — Orange flavored beverage containing erythritol

SUMMARY:
The study will determine whether acute and chronic consumption of a beverage containing erythritol will improve endothelial function in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Otherwise healthy

Exclusion Criteria:

* Pregnant
* BMI>35 kg/m2
* Long acting insulin treatment
* Other major illness, drug abuse
* Treatment with an investigational drug within 12 weeks
* Treatment with dietary or vitamin supplements
* Smoking within 3 months

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow mediated dilation | Change from baseline at 28 days

SECONDARY OUTCOMES:
Brachial artery flow-mediated dilation | Change from baseline at 2 hours
  Reactive hyperemia, carotid femoral pulse wave velocity, fingertip tonometry.
Reactive hyperemia | Change from baseline at 2 hours and 28 days
Carotid femoral pulse wave velocity | Change from baseline at 28 days
Fingertip tonometry | Change from baseline at 2 hours and 28 days
Urine F2 isoprostanes | Change from baseline at 28 days
C-reactive protein | Change from baseline at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Vita, MD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Flint N, Hamburg NM, Holbrook M, Dorsey PG, LeLeiko RM, Berger A, de Cock P, Bosscher D, Vita JA. Effects of erythritol on endothelial function in patients with type 2 diabetes mellitus: a pilot study. Acta Diabetol. 2014;51(3):513-6. doi: 10.1007/s00592-013-0534-2. Epub 2013 Dec 24. PMID 24366423